CLINICAL TRIAL: NCT07038408
Title: Multi-center, Open-label, Prospective, Randomized Study to Show Long-term Efficacy of DCB Treatment With Bail-out BRS in Comparison to BRS Treatment of De-novo Native Coronary Artery Lesions in a Relatively Young PCI Population.
Brief Title: Leave Nothing Behind Study Which Compares DCB With Bail Out BRS Versus BRS Strategy Alone
Acronym: LNB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceric Sàrl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Leave Nothing Behind
Record Dates: First submitted 2025-06-06; First posted 2025-06-26 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Drug Coated Balloon; Bioresorbable Scaffold; Percutaneous Coronary Intervention (PCI); Acute Coronary Syndrome (ACS)
Keywords: MULTI-CENTER; OPEN-LABEL; PROSPECTIVE; RANDOMIZED STUDY; LONG-TERM EFFICACY OF DCB TREATMENT WITH BAIL-OUT BRS; BRS TREATMENT; DE-NOVO NATIVE CORONARY ARTERY LESIONS; YOUNG PCI POPULATION
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB treatment (Mozec SEB) (Experimental): Mozec SEB is used during the angioplasty (V2) for patients randomized in the DCB arm with bail-out BRS. If the operator considers the results as insufficient, the MeRes100 is also used in the patient.
  Interventions: Procedure: Angioplasty with DCB (bail-out BRS)
- BRS treatment (MeRes100) (Active Comparator): MeRes100 is used during the angioplasty (V2) for patients randomized in the BRS arm.
  Interventions: Procedure: Angioplasty with DCB (bail-out BRS); Procedure: Angioplasty with BRS

INTERVENTIONS:
Procedure: Angioplasty with DCB (bail-out BRS) — Angioplasty starts with lesion preparation in both arms with a PTCA balloon catheter.
  The lesion is treated with the Mozec SEB through femoral or brachial artery. The DCB should be delivered to the target lesion within 120 seconds of insertion into the guide catheter. Under fluoroscopic visualization, the DCB is inflated at least 30 seconds (single inflation). If the results are insufficient, multiple inflation is permitted. If despite appropriate delivery and inflation of the DCB, the results remain insufficient bail-out BRS should be performed.
  Bail-out BRS is performed through femoral or brachial artery. After correct positioning, the BRS is deployed slowly, i.e. 10 seconds/atm up to 4 atm, then 5 seconds/atm up to nominal pressure or higher until desired expansion is obtained. After desired expansion obtained, pressure is maintained for 30 seconds before balloon deflation. After BRS implantation, Optical Coherence Tomography (OCT) is performed, if available.
  Other Names: DCB arm with bail-out BRS
Procedure: Angioplasty with BRS — Bail-out BRS is performed through femoral or brachial artery. BRS implantation is guided by OCT, if available. After correct positioning, the BRS is deployed slowly, i.e. 10 seconds/atm up to 4 atm, then 5 seconds/atm up to nominal pressure or higher until desired expansion is obtained. After desired expansion obtained, pressure is maintained for 30 seconds before balloon deflation. After BRS implantation, OCT is performed, if available.
  Other Names: BRS arm
  Arms: BRS treatment (MeRes100)

SUMMARY:
The goal of this study is to investigate the equivalence in early and long-term efficacy between the two "Leave nothing behind strategies" (Drug-Coated Baloon [DCB] strategy with bail-out BioResorbable Scaffold [BRS] versus BRS strategy) of de-novo native coronary artery lesions in a relatively young Percutaneous Coronary Intervention (PCI) population, to be more specific, Patients with Chronic Coronary Syndromes (CCS) and Acute Coronary Syndrome (ACS) (Non-ST-segment Elevation Myocardial Infarction [NSTEMI] and Unstable angina) between 18-68 years of age scheduled for PCI. The main questions aim to answer are:

DCB strategy with bail-out BRS implantation has equivalent clinical outcomes at 12 months compared to BRS strategy? DCB strategy with bail-out BRS implantation has noninferior angiographic in-segment net gain at 13 months compared to BRS strategy? DCB strategy with bail-out BRS implantation has equivalent clinical outcomes at 60 months compared to BRS strategy?

Participants will be followed at:

1. st FU visit - 1 month (in hospital)
2. nd FU visit - 6 months (telephone)
3. rd FU visit - 365 days±15 days (telephone) - 1Y Primary efficacy endpoint
4. th FU visit - 395 days±15 days (in hospital) co-primary efficacy endpoint for the angiographic substudy
5. th FU visit - 730 days±30 days (telephone call) - 2Y
6. th FU visit - 1095 days±30 days (telephone call) - 3Y
7. th FU visit - 1460 days±30 days (telephone call) - 4Y
8. th FU visit- 1825 days±30 days (telephone call) - 5Y

DETAILED DESCRIPTION:
The Leave Nothing Behind Study is an is an investigator-initiated trial. The Primary efficacy endpoint is target-vessel failure (TVF), defined as the composite of cardiovascular death, target-vessel myocardial infarction or ischemia-driven target-vessel revascularization (TVR) at 12 months.

Co-primary efficacy endpoint (angiographic substudy) is the in-segment net gain at 13 months.

Investigators aim to enroll 2256 patients in the main study and 196 patients in the angiographic substudy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years ≤ 68 years
* Single vessel or multivessel disease with low to moderate complex de-novo native coronary artery lesions up to 30 mm length and reference vessel diameter 2.75-4.0 mm
* Maximum of 3 target lesions
* Maximal cumulative lesion length of all treated lesions 80 mm
* Signed informed consent for participation in the study

Exclusion Criteria:

* ST-segment Elevation Myocardial Infarction (STEMI) treatment at index or in the previous 48 hours
* Severe calcified lesions
* Bifurcations lesions with planned 2 device strategy
* Left-Main (LM) disease ≥ 50% diameter stenosis
* More than 3 target lesions
* Renal insufficiency with Glomerular Filtration Rate (GFR) < 45 ml/min
* Life expectancy less than 1 year
* Known hypersensitivity or allergy to aspirin or P2Y12 receptor inhibitors
* Incapable of providing written informed consent
* Pregnant or breastfeeding women
* Under judicial protection, tutorship, or curatorship
* Participation in another trial

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2256 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-02-20 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Target-vessel Failure (TVF) | From enrollment to the end of treatment at 12 months
  Target vessel failiure is defined as the composite of cardiovascular death, target-vessel myocardial infarction or ischemia-driven target-vessel revascularization

SECONDARY OUTCOMES:
Target-Vessel Failure (TVF) at 2, 3, 4 and 5 years. | From enrollment to the end of treatment at every year from 2 years until 5 years follow-up
  Target vessel failiure is defined as the composite of cardiovascular death, target-vessel myocardial infarction or ischemia-driven target-vessel revascularization
Target-Lesion Failure (TLF) | From enrollment to the end of treatment every year until end of 5 years
  Target Lesion Failure is is defined as the composite of cardiac death, target vessel-related myocardial infarction (Q wave and non-Q wave) and ischemia-driven target lesion revascularization
(Bleeding Academic Research Consortium) BARC 2, 3 or 5 bleedings | From enrollment to the end of treatment every year until end of 5 years
  BARC definitions Type 2: any overt, actionable sign of hemorrhage that does not fit the criteria for type 3, type 4, or type 5 but does meet at least one of the following criteria: requiring nonsurgical, medical intervention by a health care professional; leading to hospitalization or increased level of care; or prompting evaluation.
  Type 3a: overt bleeding plus a hemoglobin drop of 3 to 5 g/dL* ; any transfusion with overt bleeding.
  Type 3b: overt bleeding plus a hemoglobin drop of 5 g/dL ; cardiac tamponade; bleeding requiring surgical intervention for control ; bleeding requiring intravenous vasoactive agens.
  Type 3c: intracranial hemorrhage
Net Adverse Clinical Event (NACE) | From enrollment to the end of treatment every year until end of 5 years
  NACE defined as all-cause death, myocardial infarction, all-stroke, ischemia driven TVR or BARC 3 or 5 bleeding

OTHER OUTCOMES:
Acute Gain | From enrollment to the end of treatment at 13 months
  Acute gain (in-lesion and in-segment)
Late Loss | From enrollment to the end of treatment at 13 months
  Late loss (in-lesion and in-segment)
In-segment Late Lumen Loss (LLL) | From enrollment to the end of treatment at 13 months
  In segment LLL in vessels with RVD < 3.0 mm and ≥ 3.0 mm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verma PK, Sroa S, Koushal P. A real-world experience with a thin-strut bioresorbable vascular scaffold system: a single-centre study. AsiaIntervention. 2025 Mar 20;11(1):26-34. doi: 10.4244/AIJ-D-24-00033. eCollection 2025 Mar. PMID 40114731
- [Background] Abizaid A, Kedev S, Ali RBM, Santoso T, Cequier A, van Geuns RVG, Chevalier B, Hellig F, Costa R, Onuma Y, Costa JR Jr, Serruys P, Bangalore S. Imaging and 2-year clinical outcomes of thin strut sirolimus-eluting bioresorbable vascular scaffold: The MeRes-1 extend trial. Catheter Cardiovasc Interv. 2021 Nov 15;98(6):1102-1110. doi: 10.1002/ccd.29396. Epub 2020 Dec 2. PMID 33269506
- [Background] Seth A, Onuma Y, Chandra P, Bahl VK, Manjunath CN, Mahajan AU, Kumar V, Goel PK, Wander GS, Kaul U, Ajit Kumar VK, Abizaid A, Serruys PW. Three-year clinical and two-year multimodality imaging outcomes of a thin-strut sirolimus-eluting bioresorbable vascular scaffold: MeRes-1 trial. EuroIntervention. 2019 Sep 20;15(7):607-614. doi: 10.4244/EIJ-D-19-00324. PMID 31147308
- [Background] Premchand Jain RK, Parikh K, Sethuraman S, Sharma K, Roy S, Vithala SR, Gollamandala KR, Packirisamy G, Mantravadi SS, Roleder T. Safety and Performance of the MOZEC Sirolimus-Eluting Coronary Balloon in the Treatment of Stenotic Coronary Artery Lesions: A Real-World, Multicenter, Post-Marketing Surveillance Study. Cardiol Res. 2025 Apr;16(2):130-139. doi: 10.14740/cr2026. Epub 2025 Feb 28. PMID 40051667
- [Background] Capodanno D, Angiolillo DJ. Antiplatelet Therapy After Implantation of Bioresorbable Vascular Scaffolds: A Review of the Published Data, Practical Recommendations, and Future Directions. JACC Cardiovasc Interv. 2017 Mar 13;10(5):425-437. doi: 10.1016/j.jcin.2016.12.279. PMID 28279311
- [Background] Tamburino C, Latib A, van Geuns RJ, Sabate M, Mehilli J, Gori T, Achenbach S, Alvarez MP, Nef H, Lesiak M, Di Mario C, Colombo A, Naber CK, Caramanno G, Capranzano P, Brugaletta S, Geraci S, Araszkiewicz A, Mattesini A, Pyxaras SA, Rzeszutko L, Depukat R, Diletti R, Boone E, Capodanno D, Dudek D. Contemporary practice and technical aspects in coronary intervention with bioresorbable scaffolds: a European perspective. EuroIntervention. 2015 May;11(1):45-52. doi: 10.4244/EIJY15M01_05. PMID 25599676
- [Background] Vanoverbeke L, Bennett J. Drug-eluting resorbable coronary scaffolds: a review of recent advances. Expert Opin Drug Deliv. 2025 Jul;22(7):919-933. doi: 10.1080/17425247.2025.2495043. Epub 2025 Apr 20. PMID 40238640
- [Background] Power DA, Camaj A, Kereiakes DJ, Ellis SG, Gao R, Kimura T, Ali ZA, Stockelman KA, Dressler O, Onuma Y, Serruys PW, Stone GW; ABSORB Investigators. Early and Late Outcomes With the Absorb Bioresorbable Vascular Scaffold: Final Report From the ABSORB Clinical Trial Program. JACC Cardiovasc Interv. 2025 Jan 13;18(1):1-11. doi: 10.1016/j.jcin.2024.08.050. PMID 39814482
- [Background] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887
- [Background] Stefanini GG, Holmes DR Jr. Drug-eluting coronary-artery stents. N Engl J Med. 2013 Jan 17;368(3):254-65. doi: 10.1056/NEJMra1210816. No abstract available. PMID 23323902
- [Background] Zhang YJ, Bourantas CV, Muramatsu T, Iqbal J, Farooq V, Diletti R, Campos CA, Onuma Y, Garcia-Garcia HM, Serruys PW. Comparison of acute gain and late lumen loss after PCI with bioresorbable vascular scaffolds versus everolimus-eluting stents: an exploratory observational study prior to a randomised trial. EuroIntervention. 2014 Oct;10(6):672-80. doi: 10.4244/EIJV10I6A118. PMID 24472767
- [Background] Asano T, Serruys PW, Collet C, Miyazaki Y, Takahashi K, Chichareon P, Katagiri Y, Modolo R, Tenekecioglu E, Morel MA, Garg S, Wykrzykowska J, Piek JJ, Sabate M, Morice MC, Chevalier B, Windecker S, Onuma Y. Angiographic late lumen loss revisited: impact on long-term target lesion revascularization. Eur Heart J. 2018 Sep 21;39(36):3381-3389. doi: 10.1093/eurheartj/ehy436. PMID 30124834
- [Background] Madhavan MV, Kirtane AJ, Redfors B, Genereux P, Ben-Yehuda O, Palmerini T, Benedetto U, Biondi-Zoccai G, Smits PC, von Birgelen C, Mehran R, McAndrew T, Serruys PW, Leon MB, Pocock SJ, Stone GW. Stent-Related Adverse Events >1 Year After Percutaneous Coronary Intervention. J Am Coll Cardiol. 2020 Feb 18;75(6):590-604. doi: 10.1016/j.jacc.2019.11.058. PMID 32057373